CLINICAL TRIAL: NCT05776745
Title: Study of Speech Function in Epileptic Patients Based on Stereoelectroencephalography Signal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Hemmings Wu, Neurosurgeon, Assistant Professor, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-0113
Record Dates: First submitted 2023-02-07; First posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Epilepsy
Keywords: Epilepsy; Stereoelectroencephalography; Speech
MeSH Terms: conditions — Epilepsy; Speech

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Epileptic (Experimental): Epileptic with stereoelectroencephalography
  Interventions: Behavioral: Speech; Device: Stereoelectroencephalography

INTERVENTIONS:
Behavioral: Speech — Patients read specific words and sentences
Device: Stereoelectroencephalography — Using stereoelectroencephalography to record the Intracranial EEG of the patient

SUMMARY:
Based on stereoelectroencephalography model in the treatment of epilepsy patients, this study conducted language-related experimental studies without interfering with normal monitoring treatment. Meanwhile, voice data and intracranial electrophysiological data were collected for analysis. To study the mechanism related to the language function of patients, try to establish a model to decode the intracranial electrophysiological data related to language.

ELIGIBILITY:
Inclusion Criteria:

* Patients with focal refractory epilepsy also need preoperative evaluation with SEEG

Exclusion Criteria:

* History of major depression or psychiatric disorders and medication that causes symptoms of psychiatric disorders
* Patients with severe cognitive impairment (MMSE score ≤15), unable to complete the language function test

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2022-03-20 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2023-12-25 (Estimated)

PRIMARY OUTCOMES:
Phonetic Feature Encoding in Human Superior Temporal Gyrus | through study completion, an average of 1 year
  Phonetic Feature Encoding in Human Superior Temporal Gyrus

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang University School of Medicine Second Affiliated Hospital, Hangzhou, Zhejiang, China